CLINICAL TRIAL: NCT05635279
Title: Study on the Effect of Nutritional Indices on the Prognosis of Hepatocellular Carcinoma Patients
Brief Title: Effect of Nutritional Indices on the Prognosis of HCC Patients
Status: Completed | Type: Observational
Sponsor: Juan Kang (Other)
Responsible Party: Sponsor-Investigator, Juan Kang, associate professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2022-182
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: prognostic nutritional index; psoas muscle index; geriatric nutritional risk index; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HCC patients who received ICIs combined with TKIs: HCC patients who received ICIs combined with TKIs regularly and periodically.
- HCC patients treated with TACE: HCC patients who underwent TACE as initial treatment.

INTERVENTIONS:
Other:

SUMMARY:
Primary liver cancer has recently ranked among the leading causes of cancer death, with hepatocellular carcinoma (HCC) accounting for 75%-85% of these cases. In recent years, immune checkpoint inhibitors (ICIs) combined with tyrosine kinase inhibitors (TKIs) have achieved good results in the treatment of advanced HCC patients. So far, there is a lack of studies exploring the relationship between nutritional index and the prognosis of HCC patients treated with ICIs combined with TKIs, and there are few studies on the prognostic value of nutritional index in HCC patients treated with transarterial chemoembolization (TACE). This retrospective study aims to analyze the prognostic value of prognostic nutritional index(PNI)，body mass index (BMI), psoas muscle index（PMI）and geriatric nutritional risk index (GNRI) in HCC patients who received ICIs combined with TKIs or TACE, and to provide reference for the selection of nutritional intervention programs for HCC patients.

DETAILED DESCRIPTION:
Patients who confirmed HCC in the Second Affiliated Hospital of Chongqing Medical University were enrolled in the retrospective study. The subjects were divided into two cohorts, both of which met the inclusion and exclusion criteria.The data needed to be collected included age, gender, height and weight at initial treatment and regular follow-up. Blood routine, liver function, kidney function, coagulation function, electrolytes, PIVKA-II, AFP, HBV-DNA, CT, MRI information, China liver cancer staging (CNLC), complications, treatment plan, etc. Follow-up time after initiation of treatment and time of death or significant disease progression. The survival was estimated by the Kaplan-Meier method and curves were compared by the log-rank test.Logistic regression was used to univariate and multivariate analyze the effect of variables on the outcome. Variables with P<0.05 on a univariate analysis were subjected to a multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:HCC patients received ICIs combined with TKIs regularly and periodically.

Cohort 2:HCC patients who underwent TACE as initial treatment.

Exclusion Criteria:

1. Patients with systemic malignant tumors other than HCC.
2. Patients with severe hypertension, diabetes, coronary heart disease, systemic infection and other serious diseases.
3. patients with immunodeficiency or autoimmune diseases.
4. Patients with severe malnutrition.
5. Not adhering to regular and periodic treatment.
6. Patients without regular follow-up or with missing data to be collected.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who confirmed HCC in the Second Affiliated Hospital of Chongqing Medical University were enrolled in the retrospective study. The subjects were divided into two cohorts, both of which met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Death | November 2022 to May 2024
  Death due to hepatocellular carcinoma progression

SECONDARY OUTCOMES:
Censored | November 2022 to May 2024
  Death due to other causes such as car accidents or loss to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Juan Kang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Luo N, Li H, Luo Y, Hu P, Liang L, Zhang R, Zhang D, Cai D, Kang J. Prognostic significance of psoas muscle index in male hepatocellular carcinoma patients treated with immune checkpoint inhibitors and tyrosine kinase inhibitors. Hum Vaccin Immunother. 2023 Aug;19(2):2258567. doi: 10.1080/21645515.2023.2258567. Epub 2023 Sep 20. PMID 37728115